CLINICAL TRIAL: NCT07111208
Title: Noise and/or Ultrafine Particulate Matter Induced Cerebral and Cardiovascular Damage: Experimental and Epidemiological Studies (MARKOPOLO) and Lifestyle Intervention to Attenuate Cardiovascular Health Risk (METSGREEN)
Brief Title: Ambient Air and Noise Effect on Cardiovascular Health Risk and Lifestyle Intervention to Attenuate It (METSGREEN)
Acronym: METSGREEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Grazuleviciene (Other)
Collaborators: Lithuanian University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Regina Grazuleviciene, professor, Vytautas Magnus University
Organization: Vytautas Magnus University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-07-03 No. BE-2-43; 101156161 (Other Grant/Funding Number: EU HORIZON-CL1-2024-ENVHLTH-02-06-two-stage)
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases (CVD); Metabolic Syndrome; Air Pollution Exposure; Environmental Exposure; Health Behavior Change
Keywords: ultrafine particles; noise pollution; cardiovascular risk; metabolic syndrome; physical activity; Mediterranean diet; environmental exposure
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (usual routine) (No Intervention): Participants in this group will continue their regular daily activities without any changes imposed. They will not receive specific instructions on physical activity or diet but will undergo the same measurements and monitoring as other groups for comparison purposes.
- Green Space Activity Group - Daily Physical Activity (Experimental): Participants in this group will be instructed to take a brisk 30-minute walk each day in designated urban green spaces (e.g., parks, forested areas). Physical activity will be monitored using Fitbit Alta wristband sensors to track duration, intensity, and steps.
  Interventions: Behavioral: Green Space Activity Group - Daily Physical Activity
- Mediterranean Diet Group - Dietary Intervention (Experimental): Participants in this group will follow the principles of the Mediterranean diet, including increased consumption of fruits, vegetables, whole grains, legumes, nuts, and olive oil, and reduced intake of red meat and processed foods. They will receive dietary guidance and support for meal planning throughout the 7-day intervention.
  Interventions: Behavioral: Mediterranean Diet Group - Dietary Intervention

INTERVENTIONS:
Behavioral: Green Space Activity Group - Daily Physical Activity — Participants in this group will be instructed to take a brisk 30-minute walk each day in designated urban green spaces (e.g., parks, forested areas). Physical activity will be monitored using Fitbit Alta wristband sensors to track duration, intensity, and steps.
  Arms: Green Space Activity Group - Daily Physical Activity
Behavioral: Mediterranean Diet Group - Dietary Intervention — Participants in this group will follow the principles of the Mediterranean diet, including increased consumption of fruits, vegetables, whole grains, legumes, nuts, and olive oil, and reduced intake of red meat and processed foods. They will receive dietary guidance and support for meal planning throughout the 7-day intervention.
  Arms: Mediterranean Diet Group - Dietary Intervention

SUMMARY:
This study, combining both an observational study and an interventional clinical trial, aims to assess how exposure to ultrafine particulate matter (PM0.1) and noise pollution affects the risk of cardiovascular diseases and metabolic disorders in 45-64-year-old residents of Kaunas City, and whether lifestyle interventions-specifically physical activity in green spaces and the Mediterranean diet-can help reduce these risks.

In the observational part, approximately 1,000 randomly selected 45-64 years men and women living in private households will complete an anonymous online health and lifestyle questionnaire. The clinical interventional trial will include 180 participants, who agreed to participate in the clinical study and, who meet specific health criteria. The main questions the study seeks to answer are: whether increased exposure to PM0.1 and noise is linked to higher cardiovascular and metabolic risk; and whether short-term healthy lifestyle changes can improve biological markers associated with these conditions.

Participants in the clinical trial will be randomly assigned to one of three groups: (1) control group continuing usual habits, (2) physical activity group at least 30-minute daily walks in green spaces, or (3) group adherence to a Mediterranean diet. They will have two visits to the clinic for health surveys:

* Wear a wristband sensor for 7 days to monitor physical activity, heart rate, and sleep quality
* Visit a clinic on Day 1 and Day 8 for measurements (blood pressure, waist circumference, body composition) and give blood samples for biomarker analysis.

This research will provide new evidence on environmental health risks and practical recommendations for reducing the burden of metabolic and cardiovascular diseases.

DETAILED DESCRIPTION:
The METSGREEN study is a hybrid biomedical research project combining an observational environmental-epidemiological study with an experimental clinical trial of healthy behavior. It is implemented under the international MARKOPOLO project framework, funded by the European Commission through the Horizon Europe program. The study is led in Lithuania by Vytautas Magnus University (VMU), with contributions from 15 academic institutions across Europe and North America. METSGREEN aims to explore the impact of ultrafine particulate matter (PM0.1) and noise exposure on cardiometabolic health in middle-aged urban populations and assess whether targeted lifestyle interventions can mitigate these effects.

Scientific Background and Rationale: Environmental pollution is increasingly recognized as a major contributor to chronic non-communicable diseases. Ultrafine particles (diameter <0.1 µm) are especially harmful due to their ability to penetrate deep into the respiratory tract, cross alveolar membranes, and enter systemic circulation. These particles trigger oxidative stress, systemic inflammation, endothelial dysfunction, and coagulation disorder processes implicated in the pathogenesis of metabolic syndrome and cardiovascular diseases (CVD). Epidemiological studies suggest a strong link between long-term exposure to PM0.1 and increased incidence of hypertension, diabetes, central obesity, and other metabolic risk factors. Moreover, urban noise exposure has been shown to exacerbate cardiovascular risks through stress-mediated neuroendocrine pathways. However, many of these associations remain insufficiently understood, particularly in populations with specific vulnerabilities, such as older age or lower socioeconomic status.

Nature-based interventions such as physical activity in green spaces are a promising strategy to counteract these effects. Regular exposure to nature has been shown to improve autonomic nervous system balance, reduce cortisol levels, and promote cardiovascular resilience. Dietary interventions, particularly the Mediterranean diet, rich in unsaturated fats, antioxidants, and anti-inflammatory nutrients, are also recognized for their cardioprotective effects. Despite this, very few studies integrate objective environmental exposure assessments with clinical lifestyle interventions and biomarker-based outcomes.

Study Objectives: The study is divided into two core components with distinct but complementary objectives:

1. Observational Study (n = 1,000): Model and map environmental exposure to PM0.1 and noise across Kaunas city using land-use regression (LUR) based on data collected at 20 strategic locations. Link environmental exposure estimates to self-reported health status, lifestyle factors, and socioeconomic characteristics using a standardized, anonymized online questionnaire. Assess associations between PM0.1/noise exposure and key cardiometabolic indicators: prevalence of cardiovascular disease, blood pressure, waist circumference, and anthropometric data. Investigate potential effect modifiers such as sex, age, residential environment, and economic status.
2. Experimental Clinical Trial (n = 180): Assess the short-term impact of a healthy lifestyle intervention on metabolic health indicators and biological markers in individuals with early signs of metabolic syndrome (central obesity and/or elevated blood pressure). Compare three groups (1:1:1 allocation): control (no intervention), physical activity in green space (daily 30-minute brisk walk), and Mediterranean diet intervention (dietary counselling and meal planning). Evaluate changes in biological markers (HDL, triglycerides, fasting glucose, body composition, blood pressure, etc.) and omics-level indicators (metabolomics, proteomics, DNA methylation). Determine the interaction between environmental exposure levels and response to lifestyle changes.

Study Population: Participants in the observational component are Kaunas city residents aged 45-64, randomly selected from residential registries, excluding individuals in institutional care. The clinical trial cohort will be drawn from this group and include only those with signs of metabolic disturbance, stable health status, and willingness to participate in daily monitoring and clinical visits. Exclusion criteria include pregnancy, severe cardiovascular or neurological disease, alcohol dependence, limited mobility, and use of pacemakers.

Intervention Protocol: Participants in the intervention arms will be instructed to follow specific behavioral guidelines over a 7-day period. Green Space Group: Perform daily 30-minute brisk walks in designated urban green areas. Compliance will be tracked via Fitbit Alta wristband sensors. Mediterranean Diet Group: Receive dietary counselling and guidance on meal preparation using approved Mediterranean food groups. Nutritional intake will be self-reported and supervised via regular communication with a dietitian. Control Group: Continue routine daily habits with no behavioral change. All participants will undergo two clinical assessments-on Day 1 and Day 8-at the Family Medicine Clinic of Kaunas Clinics. Clinical procedures include anthropometric measurements (waist circumference, body weight, height), blood pressure assessment, body composition analysis (using bioelectrical impedance), and venous blood sampling (up to 20 ml per visit). Biomarker Analysis: Collected blood samples will be analyzed for: Metabolic Indicators: Fasting plasma glucose, triglycerides, HDL cholesterol. Inflammatory Markers: Selected cytokines and proteins via immunoblotting. Advanced Omics Profiling: Targeted metabolomic, proteomic, and epigenetic analysis. Samples will be processed and analyzed at partner institutions: DNA methylation: National Center of Pathology (Lithuania), Laboratoire National de Santé (Luxembourg). Proteomics: University of Southern Denmark. Metabolomics: University of Eastern Finland.

Data Collection and Management: The study employs multiple layers of data protection, including participant coding, restricted data access, and secure storage. Online questionnaires are encrypted and anonymized. Wristband-collected data will be uploaded to a secure digital platform and linked with individual exposure estimates.

All clinical, lifestyle, and environmental data will be integrated for comprehensive statistical analysis. Multivariate logistic regression models will be applied, adjusting for potential confounders (age, gender, SES). Exposure-response relationships will be quantified using both linear and non-linear regression methods. The 99.9% confidence level and power of 80% will be maintained to minimize Type I and II errors.

Expected Outcomes: The study is expected to yield: Detailed mapping of urban PM0.1 and noise exposure across Kaunas. Quantified links between environmental exposure and cardiometabolic health. Evidence on the effectiveness of nature-based and dietary interventions in reducing metabolic disorder risk. Biomarker-based insight into pathophysiological pathways influenced by environmental stressors and lifestyle. Recommendations for local and European Union (EU) level public health strategies.

Ethical Considerations: The study has received ethical approval from the Kaunas Regional Biomedical Research Ethics Committee. Participation is voluntary, with informed consent required for the clinical trial. Participants may withdraw at any time. Minimal risks are anticipated, limited to standard blood sampling.

Data Protection: All data are handled according to the General Data Protection Regulation (GDPR). Personally identifiable data are stored separately and securely, accessible only to the principal investigator and designated team members. Participants have the right to access, correct, or withdraw their data.

Study Timeline and Dissemination: The total study duration is 48 months. Results will be published in peer-reviewed journals, presented at international conferences, and submitted to the European Environment Agency to provide evidence-based health guidelines. Lay summaries will be provided for participants and the general public.

The METSGREEN study represents an integrative approach to understanding and mitigating environmental health risks. By linking advanced exposure modelling with clinical and molecular endpoints, it aims to provide robust scientific evidence for targeted, sustainable, and preventive health strategies in urban settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-64 years
* Residence in Kaunas City
* Presence of metabolic disorder indicators (e.g., increased waist circumference and/or elevated blood pressure)
* Willingness to participate and provide written informed consent
* Agreement to wear a wristband sensor continuously for 7 days

Exclusion Criteria:

* Unstable angina or cardiomyopathy
* Blood pressure >160/110 mmHg
* Neurological diseases or limited mobility
* Presence of a cardiac pacemaker
* Pregnancy
* Alcohol dependence

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiovascular diseases (CVD) | Baseline and 12 months.
  Assessed using standardized questionnaire; Unit: % of participants with diagnosed CVD.
Blood pressure levels | Baseline and 12 months.
  measured with automated sphygmomanometer; Unit: mmHg (systolic and diastolic).
Waist circumference | Baseline and 12 months.
  measured with standard measuring tape. Unit: cm.
Anthropometric measurements (BMI) | Baseline and 12 months.
  Body Mass Index (BMI) calculated by dividing weight in kilograms by the square of height in meters (kg/m²) Measured using a calibrated scale and stadiometer; Unit: kg/m²

SECONDARY OUTCOMES:
Waist circumference | Baseline and after 7-day lifestyle intervention.
  Measured with standard measuring tape; Unit: cm
Blood pressure levels | Baseline and after 7-day lifestyle intervention
  Measured with automated sphygmomanometer; Unit: mmHg (systolic and diastolic).
High-density lipoprotein (HDL) | Baseline and after 7-day lifestyle intervention.
  measured from fasting blood samples using standard biochemical assay; Unit: mmol/L
Triglycerides | Baseline and after 7-day lifestyle intervention.
  measured from fasting blood samples using standard biochemical assay; Unit: mmol/L.
Plasma glucose | Baseline and after 7-day lifestyle intervention.
  measured from fasting blood samples using glucose oxidase method; Unit: mmol/L.
Biological markers from metabolomics, proteomics, and DNA methylation | through study completion, an average of 3 years.
  Assessed from blood samples using high-throughput omics technologies; Unit: relative expression levels (arbitrary units).

CONTACTS AND LOCATIONS:
Overall Officials: Regina Grazuleviciene, prof., Principal Investigator — Vytautas Magnus University
Locations (2):
- Lithuania (2):
  - Vytautas Magnus university, faculty of Natural Sciences, Environmental sciences, Kaunas, Kaunas County
  - Department of Family Medicine, Lithuanian University of Health Sciences, Kaunas

IPD SHARING:
Plan to Share IPD: No
Data will become available for this study and stored for 10 years after study completion at the study center. This retention period complies with international agreements to support long-term EU environmental and health programs.

REFERENCES:
- [Derived] Grazuleviciene R, Andrusaityte S, Dedele A, Kapustinskaite A. Ambient air and noise pollution effect on cardiovascular health risk and lifestyle intervention to attenuate it: study protocol for a randomized clinical trial. Front Public Health. 2026 Jan 26;14:1747963. doi: 10.3389/fpubh.2026.1747963. eCollection 2026. PMID 41668846

DOCUMENTS (2):
  • Study Protocol (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT07111208/Prot_000.pdf
  • Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT07111208/ICF_001.pdf